CLINICAL TRIAL: NCT03922490
Title: Adipose Derived Stromal Cell Transplantation as an Adjunct to Arthroscopy in Treatment of Effusion Synovitis of the Early Degenerative Knee
Brief Title: Lipogems Prospective Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment was suspended due to the COVID pandemic and it was decided not to resume the study.
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-1534
Record Dates: First submitted 2019-04-10; First posted 2019-04-22 (Actual); Results first posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Debridement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Knee Arthroscopy + Adipose Derived Stem Cells (ADSC) (Experimental): Experimental Group: will undergo diagnostic knee arthroscopy with injection of adipose derived stem cells. Will also carry out all procedures associated with study (Physical Exam, Magnetic Resonance Imaging (MRIs), X-rays, Questionnaires).
  Interventions: Device: Lipogems Device PLUS debridement
- Observation Cohort: Knee Arthroscopy (Other): Observational Group: will undergo diagnostic knee arthroscopy (No injection of adipose derived stem cells). Will also carry out all procedures associated with study (Physical Exam, MRIs, X-rays, Questionnaires).
  Interventions: Procedure: Debridement only

INTERVENTIONS:
Device: Lipogems Device PLUS debridement — Lipogems is the name of the technology used to obtain stem cells from the abdomen, which will then be injected into the knee after knee arthroscopy.
  Arms: Knee Arthroscopy + Adipose Derived Stem Cells (ADSC)
Procedure: Debridement only — Patients will undergo knee arthroscopy as a standard treatment for their condition but will not receive the fat-derived stem cell treatment nor will undergo any additional procedures.
  Arms: Observation Cohort: Knee Arthroscopy

SUMMARY:
The purpose of this study is to study the clinical outcomes and effects of the injection of fat-derived stem cells (the scientific name being "adipose derived autologous stem cell transplantation (ADAT)") as an addition to knee arthroscopy in the treatment of knee swelling and pain associated with mild to moderate knee osteoarthritis. Management of this condition remains a pervasive problem within orthopaedics. Lipogems is a Food and Drug Administration (FDA) approved technique. Lipogems is the name of the technology used to obtain stem cells from fat that will be aspirated/removed by suction from the abdomen. Fat will be processed to obtain stem cells which will then be injected into the knee after the physician completes knee arthroscopy. The study that we are asking patients to enroll in is important because it will attempt to answer the question about whether fat-derived stem cells added to knee arthroscopy is better, worse or no different than knee arthroscopy alone. Currently, without this study, we do not have an answer to this question.

DETAILED DESCRIPTION:
Protocol Outline:

* The patient will undergo a diagnostic knee arthroscopy. This procedure would have been performed regardless of enrollment in the study. During the diagnostic knee arthroscopy, the surgeon will determine whether the patient is eligible to participate in the study.
* If the patient has a torn meniscus, inflamed joint lining or loose fragments in the knee, this will be removed and treated and he/she will still be eligible for the study.
* If, however, the physician determines that the patient needs more invasive treatments (such as cartilage transplantation, meniscal repair, removal of a substantial amount of your meniscus), then he/she will be excluded from the study and will not have fat tissue suctioned from his/her abdomen. The standard of care treatment will then proceed based on the physician's judgement.
* After the surgeon completes the arthroscopic procedure, the recommended amount of fat-derived stem cells (about 2 teaspoons) will be injected into the knee. There will be approximately 1 teaspoon of excess fat derived stem cells, which will be transported to our research facility so that the contents can be stored for later examination.
* After surgery, 5 visits are required by the patient over the following 12 months: at 2 weeks after surgery to monitor his/her incision, at 6 weeks, 12 weeks, 6 months and then finally 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Knee pain and symptoms for >2 months - clicking, popping, giving way, pain with pivot or torque, pain that is episodic, and pain that is acute and localized to one joint
* Conservative treatment >4 weeks with one or more of:
* Non-steroidal Anti-inflammatory Drugs (NSAIDS) or acetaminophen or contraindication to use of NSAIDs and acetaminophen, Activity limitations, Physical Therapy (PT)
* Hospital for Special Surgery (HSS) MRI demonstrating grade 1-3 knee joint effusion/synovitis based on MRI Osteoarthritis Knee Score (MOAKS) criteria
* K-L grade 0-3 on radiographs and/or cartilage thinning on MRI w/ or w/o meniscal tear
* Ability to provide informed consent

Exclusion Criteria: The patients listed below are excluded due to potential confound factors which may alter clinical outcomes in either treatment group (1,3,4,5 7,8, 11, 12,13), if they may potentially cause a ceiling or floor effect to our clinical outcomes (2,6,) or if the treatment may constitute and undue risk to the patient or be outside of the standard of practice of treatment for that patient (1, 9, 10,14, 15, 16)

* 1. Under 18 years of age or skeletally immature
* 2. Grade 4 radiographic Osteoarthritis (OA) as defined by the K-L classification
* 3. Grade 4 chondral lesion of patellofemoral joint on diagnostic arthroscopy
* 4. Major coronal plane malalignment (>5° valgus or varus deviation)
* 5. Knee ligamentous instability
* 6. Pretreatment Numeric Rating Scale (NRS) pain score of <40 of 100
* 7. Systemic disorders such as diabetes, inflammatory arthritis (Rheumatoid Arthritis (RA), gout, psoriatic arthritis, Calcium Pyrophosphate Deposition Diseases (CPPD)), hematological diseases (coagulopathies),severe cardiovascular diseases, systemic infections, or immunodeficiencies.
* 8. History of septic arthritis
* 9. Ventral hernia (if abdominal donor site)
* 10. Lipomatous neoplasm in region of proposed donor site.
* 11. Current use of anticoagulant medications in the 5 days before surgical intervention
* 12. Recent intra-articular injection of corticosteroids (within 30 days) or
* 13. prior treatment with Hyaluronic acid (HA) in past 6 months.
* 14. Knee surgery within the previous 2 months
* 15. Pregnancy or possible pregnancy
* 16. Epilepsy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Riley Williams, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atukorala I, Kwoh CK, Guermazi A, Roemer F, Boudreau R, Hannon MJ, Hunter DJ. Response to: 'Synovitis in knee osteoarthritis: a precursor or concomitant feature?' by Zeng et al. Ann Rheum Dis. 2015 Oct;74(10):e59. doi: 10.1136/annrheumdis-2015-207800. Epub 2015 Aug 7. No abstract available. PMID 26253098
- [Background] Ceserani V, Ferri A, Berenzi A, Benetti A, Ciusani E, Pascucci L, Bazzucchi C, Cocce V, Bonomi A, Pessina A, Ghezzi E, Zeira O, Ceccarelli P, Versari S, Tremolada C, Alessandri G. Angiogenic and anti-inflammatory properties of micro-fragmented fat tissue and its derived mesenchymal stromal cells. Vasc Cell. 2016 Aug 18;8:3. doi: 10.1186/s13221-016-0037-3. eCollection 2016. PMID 27547374
- [Background] Fellows CR, Matta C, Zakany R, Khan IM, Mobasheri A. Adipose, Bone Marrow and Synovial Joint-Derived Mesenchymal Stem Cells for Cartilage Repair. Front Genet. 2016 Dec 20;7:213. doi: 10.3389/fgene.2016.00213. eCollection 2016. PMID 28066501
- [Background] Jannelli E, Fontana A. Arthroscopic treatment of chondral defects in the hip: AMIC, MACI, microfragmented adipose tissue transplantation (MATT) and other options. SICOT J. 2017;3:43. doi: 10.1051/sicotj/2017029. Epub 2017 Jun 7. PMID 28589877
- [Background] Karpinski K, Muller-Rath R, Niemeyer P, Angele P, Petersen W. Subgroups of patients with osteoarthritis and medial meniscus tear or crystal arthropathy benefit from arthroscopic treatment. Knee Surg Sports Traumatol Arthrosc. 2019 Mar;27(3):782-796. doi: 10.1007/s00167-018-5086-0. Epub 2018 Aug 20. PMID 30128683
- [Background] Koh YG, Kwon OR, Kim YS, Choi YJ, Tak DH. Adipose-Derived Mesenchymal Stem Cells With Microfracture Versus Microfracture Alone: 2-Year Follow-up of a Prospective Randomized Trial. Arthroscopy. 2016 Jan;32(1):97-109. doi: 10.1016/j.arthro.2015.09.010. Epub 2015 Nov 14. PMID 26585585
- [Background] Koh YG, Choi YJ, Kwon SK, Kim YS, Yeo JE. Clinical results and second-look arthroscopic findings after treatment with adipose-derived stem cells for knee osteoarthritis. Knee Surg Sports Traumatol Arthrosc. 2015 May;23(5):1308-1316. doi: 10.1007/s00167-013-2807-2. Epub 2013 Dec 11. PMID 24326779
- [Background] MacFarlane LA, Yang H, Collins JE, Jarraya M, Guermazi A, Mandl LA, Martin SD, Wright J, Losina E, Katz JN; MeTeOR Investigator Group. Association of Changes in Effusion-Synovitis With Progression of Cartilage Damage Over Eighteen Months in Patients With Osteoarthritis and Meniscal Tear. Arthritis Rheumatol. 2019 Jan;71(1):73-81. doi: 10.1002/art.40660. Epub 2018 Nov 29. PMID 30133187
- [Background] Marchal JA, Picon M, Peran M, Bueno C, Jimenez-Navarro M, Carrillo E, Boulaiz H, Rodriguez N, Alvarez P, Menendez P, de Teresa E, Aranega A. Purification and long-term expansion of multipotent endothelial-like cells with potential cardiovascular regeneration. Stem Cells Dev. 2012 Mar 1;21(4):562-74. doi: 10.1089/scd.2011.0072. Epub 2011 Jun 17. PMID 21542697
- [Background] Randelli P, Menon A, Ragone V, Creo P, Bergante S, Randelli F, De Girolamo L, Alfieri Montrasio U, Banfi G, Cabitza P, Tettamanti G, Anastasia L. Lipogems Product Treatment Increases the Proliferation Rate of Human Tendon Stem Cells without Affecting Their Stemness and Differentiation Capability. Stem Cells Int. 2016;2016:4373410. doi: 10.1155/2016/4373410. Epub 2016 Jan 6. PMID 27057170
- [Background] Schiavone Panni A, Vasso M, Braile A, Toro G, De Cicco A, Viggiano D, Lepore F. Preliminary results of autologous adipose-derived stem cells in early knee osteoarthritis: identification of a subpopulation with greater response. Int Orthop. 2019 Jan;43(1):7-13. doi: 10.1007/s00264-018-4182-6. Epub 2018 Oct 3. PMID 30280218
- [Background] Striano R. D., Chen H., Bilbool N., Azatullah K., Hilado J., Horan K. Case Study: Non-Responsive Knee Pain with Osteoarthritis and Concurrent Meniscal Disease Treated With Autologous Micro-Fragmented Adipose Tissue Under Continuous Ultrasound Guidance CellR4 2015; 3 (5): e1690
- [Background] Tremolada, Carlo. (2017). Mesenchymal Stem Cells and Regenerative Medicine: How Lipogems Technology Make Them Easy, Safe and More Effective to Use. MOJ Biology and Medicine. 2. 10.15406/mojbm.2017.02.00047.
- [Background] Tremolada C, Ricordi C, Caplan AI, Ventura C. Mesenchymal Stem Cells in Lipogems, a Reverse Story: from Clinical Practice to Basic Science. Methods Mol Biol. 2016;1416:109-22. doi: 10.1007/978-1-4939-3584-0_6. PMID 27236668
- [Background] Wang X, Jin X, Han W, Cao Y, Halliday A, Blizzard L, Pan F, Antony B, Cicuttini F, Jones G, Ding C. Cross-sectional and Longitudinal Associations between Knee Joint Effusion Synovitis and Knee Pain in Older Adults. J Rheumatol. 2016 Jan;43(1):121-30. doi: 10.3899/jrheum.150355. Epub 2015 Nov 15. PMID 26568597

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Knee Arthroscopy + Adipose Derived Stem Cells (ADSC) | Observation Cohort: Knee Arthroscopy
Started | 2 | 0
Completed | 0 (Due to COVID, recruiting patients was difficult and thus the study has been suspended. To add to that difficulty, RAs have not been permanent and have been leaving prior the agreed time when hired. The target number of participants was never obtained and thus the data set is incomplete.) | 0
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: Due to COVID, recruiting patients was difficult and thus the study has been suspended. To add to that difficulty, RAs have not been permanent and have been leaving prior the agreed time when hired. The target number of participants was never obtained and thus the data set is incomplete.
Groups:
- Total: Total of all reporting groups
Arm/Group | Knee Arthroscopy + Adipose Derived Stem Cells (ADSC) | Observation Cohort: Knee Arthroscopy | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants] — Population: Due to COVID, recruiting patients was difficult and thus the study has been suspended. To add to that difficulty, RAs have not been permanent and have been leaving prior the agreed time when hired. The target number of participants was never obtained and thus the data set is incomplete.
  Participants
    <=18 years | 0 |  | 0
    Between 18 and 65 years | 2 |  | 2
    >=65 years | 0 |  | 0
Age, Continuous [Mean (Full Range); unit: years] — Population: Due to COVID, recruiting patients was difficult and thus the study has been suspended. To add to that difficulty, RAs have not been permanent and have been leaving prior the agreed time when hired. The target number of participants was never obtained and thus the data set is incomplete.
  years | 56 [55 to 57] |  | 56 [55 to 57]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Due to COVID, recruiting patients was difficult and thus the study has been suspended. To add to that difficulty, RAs have not been permanent and have been leaving prior the agreed time when hired. The target number of participants was never obtained and thus the data set is incomplete.
  Participants
    Female | 1 |  | 1
    Male | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to COVID, recruiting patients was difficult and thus the study has been suspended. To add to that difficulty, RAs have not been permanent and have been leaving prior the agreed time when hired. The target number of participants was never obtained and thus the data set is incomplete.
  Participants
    Hispanic or Latino | 0 |  | 0
    Not Hispanic or Latino | 2 |  | 2
    Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants] — Population: Due to COVID, recruiting patients was difficult and thus the study has been suspended. To add to that difficulty, RAs have not been permanent and have been leaving prior the agreed time when hired. The target number of participants was never obtained and thus the data set is incomplete.
  participants
    United States | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Knee Injury and Osteoarthritis Outcome (KOOS) Pain Subscale
Description: Questions related to knee pain Scale range: 0-100 points (100 indicating no symptoms and 0 indicating extreme symptoms)
Time Frame: Baseline, 2-Week post-op, 6-Week post-op
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Knee Arthroscopy + Adipose Derived Stem Cells (ADSC) | Observation Cohort: Knee Arthroscopy
Number analyzed (Participants) | 2 | 0
score on a scale
  Baseline | 52.5 [33 to 72] |
  2-Week Post-op: number analyzed (Participants) | 1 | 0
  2-Week Post-op | 69 [69 to 69] |
  6-Week Post-op | 93 [92 to 94] |

2. Secondary Outcome: Change in Knee Injury and Osteoarthritis Outcome (KOOS) Symptoms
Description: Questions related to other knee symptoms other than pain Scale range: 0-100 points (100 indicating no symptoms and 0 indicating extreme symptoms)
Time Frame: Baseline, 2-Week post-op, 6-Week post-op
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Knee Arthroscopy + Adipose Derived Stem Cells (ADSC) | Observation Cohort: Knee Arthroscopy
Number analyzed (Participants) | 2 | 0
score on a scale
  Baseline | 51.5 [39 to 64] |
  2-Week Post-op: number analyzed (Participants) | 1 | 0
  2-Week Post-op | 75 [75 to 75] |
  6-Week Post-op | 82.5 [79 to 86] |

3. Secondary Outcome: Change in Knee Injury and Osteoarthritis Outcome (KOOS) Function in Daily Living (ADL)
Description: Questions related to function in daily living Scale range: 0-100 points (100 indicating no symptoms and 0 indicating extreme symptoms)
Time Frame: Baseline, 2-Week post-op, 6-Week post-op
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Knee Arthroscopy + Adipose Derived Stem Cells (ADSC) | Observation Cohort: Knee Arthroscopy
Number analyzed (Participants) | 2 | 0
score on a scale
  Baseline | 56 [37 to 75] |
  2-Week Post-op: number analyzed (Participants) | 1 | 0
  2-Week Post-op | 75 [75 to 75] |
  6-Week Post-op | 90.5 [87 to 94] |

4. Secondary Outcome: Change in Knee Injury and Osteoarthritis Outcome (KOOS) Function in Sport and Recreation (Sport/Rec)
Description: Questions related to function in sport and recreation Scale range: 0-100 points (100 indicating no symptoms and 0 indicating extreme symptoms)
Time Frame: Baseline, 2-Week post-op, 6-Week post-op
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Knee Arthroscopy + Adipose Derived Stem Cells (ADSC) | Observation Cohort: Knee Arthroscopy
Number analyzed (Participants) | 2 | 0
score on a scale
  Baseline | 27.5 [10 to 45] |
  2-week Post-Op: number analyzed (Participants) | 1 | 0
  2-week Post-Op | 45 [45 to 45] |
  6-Week Post-Op | 57.5 [45 to 70] |

5. Secondary Outcome: Change in Knee Injury and Osteoarthritis Outcome (KOOS) Quality of Life (QOL)
Description: Questions related to knee-related quality of life Scale range: 0-100 points (100 indicating no symptoms and 0 indicating extreme symptoms)
Time Frame: Baseline, 2-Week post-op, 6-Week post-op
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Knee Arthroscopy + Adipose Derived Stem Cells (ADSC) | Observation Cohort: Knee Arthroscopy
Number analyzed (Participants) | 2 | 0
score on a scale
  Baseline | 34.5 [19 to 50] |
  2-Week Post-op: number analyzed (Participants) | 1 | 0
  2-Week Post-op | 44 [44 to 44] |
  6-Week Post-op | 56.5 [50 to 63] |

6. Secondary Outcome: Change in International Knee Documentation Committee (IKDC) Subjective Knee Form
Description: Questions related to knee function over periods of time (100 indicating no symptoms and 0 indicating extreme symptoms)
Time Frame: Baseline, 2-Week post-op, 6-Week post-op
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Knee Arthroscopy + Adipose Derived Stem Cells (ADSC) | Observation Cohort: Knee Arthroscopy
Number analyzed (Participants) | 2 | 0
units on a scale
  Baseline | 41.4 [25.3 to 57.5] |
  2-Week Post-op: number analyzed (Participants) | 1 | 0
  2-Week Post-op | 50.6 [50.6 to 50.6] |
  6-Week Post-op | 63.8 [59.8 to 67.8] |

7. Secondary Outcome: Change in Numerical Pain Rating Scale (NPRS)
Description: Numerical pain rating scale for pain in knee (0-10) (0: no pain - 10: worst pain imaginable)
Time Frame: Baseline, 2-Week post-op, 6-Week post-op
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Knee Arthroscopy + Adipose Derived Stem Cells (ADSC) | Observation Cohort: Knee Arthroscopy
Number analyzed (Participants) | 2 | 0
score on a scale
  Baseline | 5.5 [3 to 8] |
  2-Week Post-op: number analyzed (Participants) | 1 | 0
  2-Week Post-op | 2 [2 to 2] |
  6-Week Post-op | 2.5 [2 to 3] |

8. Secondary Outcome: Change in Marx Activity Rating Scale
Description: Measures frequency of activity in healthiest and most active state during past year Includes four knee functions, each rated 0-4 total scale range 0-16 (higher score indicates more frequent participation/activity)
Time Frame: Baseline, 2-Week post-op, 6-Week post-op
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Knee Arthroscopy + Adipose Derived Stem Cells (ADSC) | Observation Cohort: Knee Arthroscopy
Number analyzed (Participants) | 2 | 0
score on a scale
  Baseline | 3.5 [0 to 7] |
  2-Week Post-op: number analyzed (Participants) | 1 | 0
  2-Week Post-op | 0 [0 to 0] |
  6-Week Post-op | 4 [0 to 8] |

9. Secondary Outcome: Change in Patient-Reported Outcomes Measurement Information System Global-10 Short Form (PROMIS-10)
Description: 10-item questionnaire with nine 5-point (as well as a single 11-point) rating scales. The results are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score". The average "T-Score" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient.
  11-point scale question recalculated to a 5 point scale. only 8 of 10 questions used for scoring calculations (Each sub-score is generated by 4/8 questions) - 4Qs, 5 points each Scale from 0-20 to calculate Global Mental Health Raw Score (higher score means better outcome) Scale from 0-20 to calculate Global Physical Health Raw Score (higher score means better outcome)
  The raw scores are then standardized to general population using the "T-score":
  Global physical health t-score range: 16.2-67.7 Global mental health t-score range: 21.2-67.6
Time Frame: Baseline, 2-Week post-op, 6-Week post-op
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: T-score
Arm/Group | Knee Arthroscopy + Adipose Derived Stem Cells (ADSC) | Observation Cohort: Knee Arthroscopy
Number analyzed (Participants) | 2 | 0
T-score
  Baseline (Global Physical Health Score) | 45 [42.3 to 47.7] |
  Baseline (Global Mental Health Score) | 52.15 [48.3 to 56] |
  2-Week Post-op (Global Physical Health Score): number analyzed (Participants) | 1 | 0
  2-Week Post-op (Global Physical Health Score) | 47.7 [47.7 to 47.7] |
  2-Week Post-op (Global Mental Health Score): number analyzed (Participants) | 1 | 0
  2-Week Post-op (Global Mental Health Score) | 56.0 [56.0 to 56.0] |
  6-Week Post-op (Global Physical Health Score) | 49.25 [47.7 to 50.8] |
  6-Week Post-Op (Global Mental Health Score) | 48.3 [48.3 to 48.3] |

ADVERSE EVENTS:
Time Frame: Up to 1 year post-op, adverse event data was collected for each patient.
Description: Due to COVID, recruiting patients was difficult and thus the study has been suspended. To add to that difficulty, RAs have not been permanent and have been leaving prior the agreed time when hired. The target number of participants was never obtained and thus the data set is incomplete.
Arm/Group | Knee Arthroscopy + Adipose Derived Stem Cells (ADSC) | Observation Cohort: Knee Arthroscopy
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0

LIMITATIONS AND CAVEATS:
Due to COVID, recruiting patients has been difficult. To add to that difficulty, RAs have not been permanent and have been leaving prior the agreed time when hired. Even though Dr. Williams prescreens patients himself for this study, without an RA it has made things much more difficult. At the moment we are in the hiring process and hope this changes for the next continuing review. There have been no changes since the last time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT03922490/Prot_002.pdf
  • Informed Consent Form (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/90/NCT03922490/ICF_003.pdf